CLINICAL TRIAL: NCT02006940
Title: Comparative Study Of The Methods Of Probe-Based Confocal Laser Endomicroscopy Of Distal Airways, High Resolution Computed Tomography And Morphology In Diagnostics Of Lung Diseases
Brief Title: The Study Of Probe-Based Confocal Laser Endomicroscopy Of Distal Airways In Diagnostics Of Lung Diseases
Acronym: pCLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FRCC FMBA
Record Dates: First submitted 2013-11-28; First posted 2013-12-10 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Inflammatory, Interstitial, Rare Lung Diseases
Keywords: alveoflex; probe-based confocal laser endomicroscopy; pCLE; alveoscopy; morphology; high resolution computed tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alveoflex, in vivo imaging miniprobe (Experimental): All the patients will be examined using confocal laser endomicroscopy during bronchoscopy with a special minirobe Alveoflex before and after the treatment. Records will be done and analyzed prospectively with the included software for endomicroscopic system.
  Interventions: Device: miniprobe Alveoflex

INTERVENTIONS:
Device: miniprobe Alveoflex — Alveoflex uses 488nm laser, generating real time moving images with an optical area of 600μm at a video frame rate of 12 images per second and a focus depth of 50μm
  Other Names: Cellvizio system (Mauna Kea Technologies, Paris, France)

SUMMARY:
The study is devoted to the comparative analysis of the data received in patients with lung pathology using new method of probe-based confocal laser endoscopy of distal airways and two reference methods: high resolution computed tomography and morphology.

DETAILED DESCRIPTION:
A relatively new technology in pulmonary medicine, probe-based confocal laser endomicroscopy of distal airways, which is also called alveoscopy, allows for real-time minimally invasive intraacinar imaging. This method has been developed that special miniprobe can be passed into the distal airway via the working channel of the bronchoscope and provide so called "optical biopsy". The method is based on the natural autofluorescence of pulmonary structures, detecting the elastin scaffold of central and peripheral airways, the structure of alveoli, blood vessels and alveolar macrophages. Taking into account the fact that in vivo endomicroscopy of distal airways is a novel diagnostic technique it needs correlating the obtained data at certain disease with the reference methods for the challenges of our current understanding of interpreting endomicroscopic images. We choose high resolution computed tomography and morphology as such reference methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed Consent;
* patients' fitness;
* the diagnosis of one of the following lung diseases: COPD, pneumonia, solitary nodule, pulmonary sarcoidosis, idiopathic interstitial pneumonia, hypersensitivity pneumonitis, pulmonary vasculitis, pulmonary eosinophilia, hemochromatosis, histiocytosis X, pulmonary lymphangioleiomyomatosis; alveolar proteinosis, other rare lung disease
* high resolution computed tomography scans performed not later than one month before pCLE;
* planned or performed histology

Exclusion Criteria:

* Severe respiratory failure,
* pregnancy or breast feeding,
* lung bleeding,
* any acute or chronic disease that may be a contraindication to bronchoscopy,
* any significant blood coagulation disorder,
* any diseases of hematopoietic system,
* alcoholism or toxic addiction,
* taking part in other clinical trials,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with the Correspondence of pCLE Images to HRCT and Morphologic Data as a Measure of Specificity and Sensitivity of the Method | up to three years
  pCLE images will be assessed morphometrically. Such criteria as quantity of alveolar macrophages, quantity of floating intraalveolar substances etc. will be measured using 6-point score, where zero means the absence of the symptom and 5 - the maximal expressiveness. Thickness of interalveolar septum, diameter of microvessels and thickness of elastic fibers will be measured using special tool with the included software for endomicroscopic system. Radiologic signs e.g. low-density areas and consolidation areas will be assessed in Hounsfield Units. Other radiologic signs e.g. ground-glass opacity, crazy paving patterns etc. will be measured by 6-point scale, the same as for pCLE images. Morphological analysis of the lung tissue specimens (received as a result of transbronchial biopsy) will be made according to the structures in pCLE images for 20 fields of view.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Olesya Danilevskaya, MD, Principal Investigator — Federal Research Clinical Center FMBA Russia
Locations (1):
- Federal Research Clinical Center FMBA Russia, Moscow, Russia

REFERENCES:
- [Derived] Danilevskaya O, Averyanov A, Lesnyak V, Chernyaev A, Sorokina A. Confocal laser endomicroscopy for diagnosis and monitoring of pulmonary alveolar proteinosis. J Bronchology Interv Pulmonol. 2015 Jan;22(1):33-40. doi: 10.1097/LBR.0000000000000126. PMID 25590481